CLINICAL TRIAL: NCT00735644
Title: Lot-to-lot Consistency, Bridging, and Safety Trial of ChimeriVax™-Japanese Encephalitis Vaccine in Toddlers in Thailand and the Philippines
Brief Title: Study of ChimeriVax™-Japanese Encephalitis Vaccine in Toddlers in Thailand and the Philippines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JEC02
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Japanese Encephalitis; Hepatitis A
Keywords: Japanese encephalitis, Hepatitis A, Inactivated Mouse-Brain
MeSH Terms: conditions — Encephalitis, Japanese; Hepatitis A | interventions — Japanese Encephalitis Vaccines; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- JE-CV GPO MBP (Lot 1) (Experimental): Participants 12 to 18 months of age received one dose of Japanese encephalitis chimeric virus vaccine (JE-CV) from Government Pharmaceutical Organization Mérieux Biological Products (GPO-MBP) Lot 1.
  Interventions: Biological: Japanese encephalitis vaccine
- JE-CV GPO MBP (Lot 2) (Experimental): Participants 12 to 18 months of age received one dose of Japanese encephalitis chimeric virus vaccine (JE-CV) from Government Pharmaceutical Organization Mérieux Biological Products (GPO-MBP) Lot 2.
  Interventions: Biological: Japanese encephalitis vaccine
- JE-CV GPO MBP (Lot 3) (Experimental): Participants 12 to 18 months of age received one dose of Japanese encephalitis chimeric virus vaccine (JE-CV) from Government Pharmaceutical Organization Mérieux Biological Products (GPO-MBP) Lot 3.
  Interventions: Biological: Japanese encephalitis vaccine
- JE-CV WRAIR (Group 4) (Active Comparator): Participants 12 to 18 months of age received one dose of JE-CV from Acambis at Walter Reed Army Institute of Research (WRAIR)
  Interventions: Biological: Japanese encephalitis vaccine (Acambis)
- Hepatitis A (Group 5) (Sham Comparator): Participants 12 to 18 months of age randomized to receive Hepatitis A vaccine
  Interventions: Biological: Hepatitis A vaccine

INTERVENTIONS:
Biological: Japanese encephalitis vaccine — 0.5 mL, Subcutaneous
  Other Names: ChimeriVax™-JE
  Arms: JE-CV GPO MBP (Lot 1)
Biological: Japanese encephalitis vaccine — 0.5 mL, Subcutaneous
  Other Names: ChimeriVax™-JE
  Arms: JE-CV GPO MBP (Lot 2)
Biological: Japanese encephalitis vaccine — 0.5 mL, Subcutaneous
  Other Names: ChimeriVax™-JE
  Arms: JE-CV GPO MBP (Lot 3)
Biological: Japanese encephalitis vaccine (Acambis) — 0.5 mL, Subcutaneous
  Arms: JE-CV WRAIR (Group 4)
Biological: Hepatitis A vaccine — 0.5 mL, Intramuscular
  Other Names: Avaxim® 80U Pediatric
  Arms: Hepatitis A (Group 5)

SUMMARY:
This study is to assess the safety and immunogenicity of three consecutive lots of JE-CV in toddlers aged 12-18 months.

Primary objective:

To demonstrate the bio-equivalence of three lots of JE-CV vaccine manufactured by sanofi pasteur.

Secondary objective:

To describe the safety of vaccination in all subjects

DETAILED DESCRIPTION:
This is a Phase III trial in toddlers in Thailand and the Philippines.

ELIGIBILITY:
Inclusion Criteria :

* Aged 12 to 18 months on the day of inclusion.
* In good general health, without significant medical history.
* Provision of informed consent form signed by at least one parent or other legally acceptable representative, and by at least one independent witness if required by local regulations.
* Subject and parent/legally acceptable representative able to attend all scheduled visits and comply with all trial procedures.
* Completion of vaccinations according to the national immunization schedule.

Exclusion Criteria :

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing any of the same substances.
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator.
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of the immune response.
* Administration of any anti-viral within 2 months preceding V01.
* History of central nervous system disorder or disease, including seizures.
* Personal or family history of thymic pathology (thymoma), thymectomy, or myasthenia.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination.
* Personal human immunodeficiency virus seropositivity in the blood sample taken at screening.
* Receipt of any JE vaccine or hepatitis A vaccine.
* Previous vaccination against flavivirus disease.
* History of flavivirus infection (confirmed either clinically, serologically or microbiologically)
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular vaccination.
* Febrile illness (temperature ≥38°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (7):
- Philippines (5):
  - Alabang
  - Bayanan
  - Buli
  - Cupang
  - Sucat
- Thailand (2):
  - Bangkok
  - Khon Kaen

REFERENCES:
- [Result] Feroldi E, Pancharoen C, Kosalaraksa P, Watanaveeradej V, Phirangkul K, Capeding MR, Boaz M, Gailhardou S, Bouckenooghe A. Single-dose, live-attenuated Japanese encephalitis vaccine in children aged 12-18 months: randomized, controlled phase 3 immunogenicity and safety trial. Hum Vaccin Immunother. 2012 Jul;8(7):929-37. doi: 10.4161/hv.20071. Epub 2012 Jul 1. PMID 22777096
- [Result] Bonaparte M, Dweik B, Feroldi E, Meric C, Bouckenooghe A, Hildreth S, Hu B, Yoksan S, Boaz M. Immune response to live-attenuated Japanese encephalitis vaccine (JE-CV) neutralizes Japanese encephalitis virus isolates from south-east Asia and India. BMC Infect Dis. 2014 Mar 21;14:156. doi: 10.1186/1471-2334-14-156. PMID 24656175
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 02 August 2008 through 27 March 2009 at 3 clinic sites in Thailand and 5 clinic sites in the Philippines.
Pre-assignment Details: A total of 1200 participants who met all of the inclusion and none of the exclusion criteria were randomized, 1199 were vaccinated in this study.
Groups:
- JE-CV GPO MBP (Lot 2): Participants 12 to 18 months of age received one dose of JE-CV from GPO MBP Lot 2
- JE-CV GPO MBP (Lot 3): Participants 12 to 18 months of age received one dose of JE- CV from GPO MBP Lot 3
- JE-CV WRAIR: Participants 12 to 18 months of age received one dose of JE-CV from Acambis at Walter Reed Army Institute of Research (WRAIR)
- Hepatitis A: Participants 12 to 18 months of age received the Hepatitis A vaccine
Period: Overall Study
Arm/Group | JE-CV GPO MBP (Lot 1) | JE-CV GPO MBP (Lot 2) | JE-CV GPO MBP (Lot 3) | JE-CV WRAIR | Hepatitis A
Started | 303 | 300 | 296 | 199 | 102
Completed | 303 | 298 | 295 | 198 | 102
Not Completed | 0 | 2 | 1 | 1 | 0
Not completed — Did not receive study vaccine | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population represents the participants who have received the trial vaccine or control vaccine (safety analysis set). Data on participants were analyzed and presented according to the vaccine they actually received.
Groups:
- JE CV GPO MBP (Lot 1): Participants 12 to 18 months of age received one dose of Japanese encephalitis chimeric virus vaccine (JE CV) from Government Pharmaceutical Organization Mérieux Biological Products (GPO MBP) Lot 1 subcutaneously
- JE-CV GPO MBP (Lot 3): Participants 12 to 18 months of age received one dose of JE-CV from GPO MBP Lot 3
- Hepatitis A: Participants 12 to 18 months of age received Hepatitis A vaccine
- Total: Total of all reporting groups
Arm/Group | JE CV GPO MBP (Lot 1) | JE-CV GPO MBP (Lot 2) | JE-CV GPO MBP (Lot 3) | JE-CV WRAIR | Hepatitis A | Total
Number analyzed (Participants) | 303 | 299 | 296 | 199 | 102 | 1199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 303 | 299 | 296 | 199 | 102 | 1199
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 14.3 (1.91) | 14.5 (1.84) | 14.4 (1.88) | 14.3 (1.81) | 14.3 (1.93) | 14.4 (1.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 138 | 143 | 94 | 45 | 575
  Male | 148 | 161 | 153 | 105 | 57 | 624
Region of Enrollment [Number; unit: Participants]
  Thailand | 123 | 122 | 121 | 82 | 42 | 490
  Philippines | 180 | 177 | 175 | 117 | 60 | 709

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroconversion to Vaccine Antigens Following Vaccination With JE-CV by GPO MBP Lots
Description: Anti-Japanese encephalitis chimeric virus vaccine antibodies were measured using the 50% plaque reduction neutralization test (PRNT50). Seroconversion was defined as participants with a pre-vaccination titer <10 1/dil and post-vaccination titer ≥ 10 1/dil, or participants with pre-vaccination titer ≥ 10 1/dil and 4-fold increase from pre- to post-vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Seroconversion to the JE CV vaccine antigens was assessed in the participants who were vaccinated and completed all study defined activities, Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | JE CV GPO MBP (Lot 1) | JE-CV GPO MBP (Lot 2) | JE-CV GPO MBP (Lot 3) | JE-CV WRAIR | Hepatitis A
Number analyzed (Participants) | 288 | 292 | 286 | 193 | 97
Participants
  JE CV Day 0 (≥10 1/dil; N=288, 290, 285, 192, 0) | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | NA [0 to 0] — Anti-Japanese encephalitis chimeric virus vaccine antibodies were not assayed in this group
  JE CV Day 28 (≥10 1/dil; N=288, 284, 283, 192, 0) | 282 | 262 [0 to 0] | 267 [0 to 0] | 185 [0 to 0] | NA [0 to 0] — Anti-Japanese encephalitis chimeric virus vaccine antibodies were not assayed in this group

2. Secondary Outcome: Geometric Mean Titers Against the Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) Antigens Before and Following Vaccination With a JE-CV by GPO MBP Lot or Walter Reed Army Institute of Research (WRAIR) JE-CV
Description: Anti-Japanese Encephalitis Chimeric Virus antibodies were measured using the 50% plaque reduction neutralization test (PRNT50) assay.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean titers against the JE CV antigens were assessed in the participants who were vaccinated and completed all study defined activities, Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | JE CV GPO MBP (Lot 1) | JE-CV GPO MBP (Lot 2) | JE-CV GPO MBP (Lot 3) | JE-CV WRAIR | Hepatitis A
Number analyzed (Participants) | 288 | 292 | 286 | 193 | 0
Titers
  Anti JE-CV Day 0 (N=288, 290, 285, 192, 0) | 5.17 [5.06 to 5.29] | 5.08 [4.99 to 5.17] | 5.19 [5.02 to 5.37] | 5.09 [4.95 to 5.24] |
  Anti JE CV Day 28 (N=288, 284, 283, 192, 0) | 212 [179 to 252] | 167 [138 to 202] | 188 [156 to 226] | 212 [168 to 268] |

3. Secondary Outcome: Number of Participants With Seroprotection to Japanese Encephalitis Chimeric Virus Antigens Before and Following Vaccination With a JE-CV by GPO MBP Lot or WRAIR JE-CV
Description: Anti-Japanese encephalitis chimeric virus vaccine antibodies were measured using the PRNT50 assay. Seroprotection was defined as the proportion of subjects with a JE CV virus PRNT50 neutralizing antibody titer ≥10 1/dilution (dil).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Seroprotection against JE CV antigens was assessed in the participants who were vaccinated and completed all study defined activities, Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Groups:
- JE-CV GPO MBP (Lot 1): Participants 12 to 18 months of age received one dose of Japanese encephalitis chimeric virus vaccine (JE-CV) from Government Pharmaceutical Organization Mérieux Biological Products (GPO MBP) Lot 1
Arm/Group | JE-CV GPO MBP (Lot 1) | JE-CV GPO MBP (Lot 2) | JE-CV GPO MBP (Lot 3) | JE-CV WRAIR | Hepatitis A
Number analyzed (Participants) | 288 | 292 | 286 | 193 | 97
Participants
  JE CV Day 0 (N=288, 290, 285, 192, 0) | 10 | 4 [0 to 0] | 8 [0 to 0] | 2 [0 to 0] | NA [0 to 0] — Japanese encephalitis chimeric virus vaccine antibodies were not measured in this group
  JE CV Day 28 (N=288, 284, 283, 192, 0) | 297 | 269 [0 to 0] | 276 [0 to 0] | 190 [0 to 0] | NA [0 to 0] — Japanese encephalitis chimeric virus vaccine antibodies were not measured in this group

4. Secondary Outcome: Geometric Mean Titers Ratios Against the Japanese Encephalitis Chimeric Virus (JE-CV) Antigen Following Vaccination With One of the JE-CV by GPO MBP Lots or WRAIR JE-CV Vaccine
Description: Anti Japanese encephalitis chimeric virus antibodies were measured using the PRNT50 assay.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean titers against the JE CV antigens were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Groups:
- JE-CV GPO MBP (Lot 1): Participants 12 to 18 months of age received one dose of Japanese encephalitis chimeric virus vaccine (JE CV) from Government Pharmaceutical Organization Mérieux Biological Products (GPO MBP) Lot 1 subcutaneously
- JE-CV MBP (Lot 2): Participants 12 to 18 months of age received one dose of JE CV from GPO MBP Lot 2 subcutaneously
- JE-CV MBP (Lot 3): Participants 12 to 18 months of age received one dose of JE CV from GPO MBP Lot 3 subcutaneously
- JE-CV WRAIR: Participants 12 to 18 months of age received one dose of JE CV from Acambis at WRAIR subcutaneously
- Hepatitis A: Participants 12 to 18 months of age received the Hepatitis vaccine intramuscularly
Arm/Group | JE-CV GPO MBP (Lot 1) | JE-CV MBP (Lot 2) | JE-CV MBP (Lot 3) | JE-CV WRAIR | Hepatitis A
Number analyzed (Participants) | 288 | 292 | 286 | 193 | 97
Titer ratio | 41.1 [34.6 to 48.7] | 32.9 [27.3 to 39.8] | 36.6 [30.3 to 44.1] | 42.2 [33.3 to 53.3] | NA [NA to NA] — Participants in this group did not receive a Japanese encephalitis chimeric virus vaccine

5. Secondary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions Following Vaccination With a Japanese Encephalitis Chimeric Virus Vaccine (JE- CV) by GPO MBP Lot or WRAIR JE-CV, or Hepatitis A Vaccine.
Description: Solicited injection site: Tenderness, Erythema, and Swelling; Solicited systemic reactions: Fever (Temperature), Vomiting, Crying Abnormal, Drowsiness, Appetite Lost, and Irritability. Grade 3 injection site: Tenderness, cries when injected limb is moved or the movement of injected limb is reduced; Erythema and Swelling ≥5 cm. Grade 3 systemic reactions: Fever, temperature >39.5˚C; Vomiting, ≥6 episodes per 24 hours or requiring parenteral hydration; Crying Abnormal, >3 hours; Drowsiness, sleeping most of the time or difficult to wake up; Appetite Lost, refuses ≥3 or most feeds/meals; and Irritability, inconsolable.
Time Frame: Day 0 up to Day 14 post-vaccination
Population: Solicited injection site and systemic reactions were assessed in the Safety Analysis Set. A participant randomized to receive JE CV GPO MBP Lot 1 vaccine, received JE CV GPO MBP Lot 3. For safety analysis, the participant was analyzed according to the actual vaccine received.
Measure: Number; unit: Participants
Arm/Group | JE CV GPO MBP (Lot 1) | JE-CV GPO MBP (Lot 2) | JE-CV GPO MBP (Lot 3) | JE-CV WRAIR | Hepatitis A
Number analyzed (Participants) | 302 | 299 | 297 | 199 | 102
Participants
  Injection site Tenderness | 58 | 59 [0 to 0] | 67 [0 to 0] | 59 [0 to 0] | 18 [0 to 0]
  Grade 3 Injection site Tenderness | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Injection site Erythema | 64 | 63 [0 to 0] | 87 [0 to 0] | 54 [0 to 0] | 26 [0 to 0]
  Grade 3 Injection site Erythema | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Injection site Swelling | 22 | 20 [0 to 0] | 21 [0 to 0] | 13 [0 to 0] | 4 [0 to 0]
  Grade 3 Injection site Swelling | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Fever | 51 | 62 [0 to 0] | 64 [0 to 0] | 48 [0 to 0] | 21 [0 to 0]
  Grade 3 Fever | 3 | 5 [0 to 0] | 3 [0 to 0] | 1 [0 to 0] | 0 [0 to 0]
  Vomiting | 60 | 57 [0 to 0] | 53 [0 to 0] | 39 [0 to 0] | 16 [0 to 0]
  Grade 3 Vomiting | 3 | 1 [0 to 0] | 1 [0 to 0] | 1 [0 to 0] | 1 [0 to 0]
  Crying Abnormal | 58 | 54 [0 to 0] | 50 [0 to 0] | 41 [0 to 0] | 21 [0 to 0]
  Grade 3 Crying Abnormal | 1 | 0 [0 to 0] | 1 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Drowsiness | 58 | 53 [0 to 0] | 53 [0 to 0] | 38 [0 to 0] | 20 [0 to 0]
  Grade 3 Drowsiness | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Appetite Lost | 82 | 71 [0 to 0] | 74 [0 to 0] | 57 [0 to 0] | 27 [0 to 0]
  Grade 3 Appetite Lost | 3 | 1 [0 to 0] | 1 [0 to 0] | 2 [0 to 0] | 0 [0 to 0]
  Irritability | 91 | 79 [0 to 0] | 79 [0 to 0] | 65 [0 to 0] | 28 [0 to 0]
  Grade 3 Irritability | 2 | 0 [0 to 0] | 1 [0 to 0] | 1 [0 to 0] | 1 [0 to 0]

6. Other Pre Specified Outcome: Serological Status of Flavivirus Infection at Baseline (Before) Vaccination With a Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) or Hepatitis A Vaccine.
Description: Flavivirus (FV) positive was defined as anti-JE against homologous virus strain ≥10 l/dil or anti dengue against at least one serotype ≥10 l/dil. FV negative was defined as anti-JE against homologous virus strain <10 l/dil and anti-dengue against the 4 serotypes <10 l/dilution.
Time Frame: Day 0 (pre-vaccination)
Population: Serological status of Flavivirus infection was assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Participants
Groups:
- JE-CV GPO MBP (Lot 1): Participants 12 to 18 months of age received one dose of Japanese encephalitis chimeric virus vaccine (JE CV) from Government Pharmaceutical Organization Mérieux Biological Products (GPO MBP) Lot 1
Arm/Group | JE-CV GPO MBP (Lot 1) | JE-CV GPO MBP (Lot 2) | JE-CV GPO MBP (Lot 3) | JE-CV WRAIR | Hepatitis A
Number analyzed (Participants) | 288 | 292 | 285 | 192 | 97
Participants
  JE CV/dengue FV positive (N=288,290,285,192,97) | 19 | 23 [0 to 0] | 32 [0 to 0] | 15 [0 to 0] | 13 [0 to 0]
  JE CV/dengue FV negative (N=288,290,285,192,97) | 265 | 266 [0 to 0] | 249 [0 to 0] | 176 [0 to 0] | 84 [0 to 0]
  JE CV (N=288, 290, 285, 192, 97) | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Dengue serotype 1 (N=284, 289, 282, 192, 97) | 17 | 19 [0 to 0] | 28 [0 to 0] | 14 [0 to 0] | 13 [0 to 0]
  Dengue serotype 2 (N=284, 289, 282, 192, 97) | 15 | 18 [0 to 0] | 26 [0 to 0] | 11 [0 to 0] | 12 [0 to 0]
  Dengue serotype 3 (N=284, 289, 282, 192, 97) | 16 | 18 [0 to 0] | 27 [0 to 0] | 12 [0 to 0] | 11 [0 to 0]
  Dengue serotype 4 (N=284, 289, 282, 192, 97) | 10 | 6 [0 to 0] | 13 [0 to 0] | 7 [0 to 0] | 8 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) data were collected from Day 0 (post-vaccination) up to Day 180 post-vaccination.
Description: The total (N) for solicited AEs in the table reflects participants for which diary cards were returned and with available data for the event during the period. A participant randomized to receive JE CV GPO MBP Lot 1 vaccine, received JE CV GPO MBP Lot 3. For safety analysis, the participant was analyzed according to the actual vaccine received.
Arm/Group | JE-CV GPO MBP (Lot 1) | JE-CV GPO MBP (Lot 2) | JE-CV GPO MBP (Lot 3) | JE-CV WRAIR | Hepatitis A
Serious Adverse Events (participants affected / at risk) | 10/302 | 17/299 | 13/297 | 7/199 | 7/102
Other Adverse Events (participants affected / at risk) | 91/302 | 99/299 | 87/297 | 65/199 | 36/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JE-CV GPO MBP (Lot 1) (N=302) | JE-CV GPO MBP (Lot 2) (N=299) | JE-CV GPO MBP (Lot 3) (N=297) | JE-CV WRAIR (N=199) | Hepatitis A (N=102)
Bronchiolitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 4 (4) | 4 (4) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 2 (2) | 6 (6) | 4 (4) | 1 (1) | 3 (4)
Amoebiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Testicular yolk sac tumour stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JE-CV GPO MBP (Lot 1) (N=302) | JE-CV GPO MBP (Lot 2) (N=299) | JE-CV GPO MBP (Lot 3) (N=297) | JE-CV WRAIR (N=199) | Hepatitis A (N=102)
Pyrexia (General disorders) | 2 (2) | 6 (6) | 6 (6) | 10 (10) | 1 (1)
Gastroenteritis (Infections and infestations) | 19 (21) | 18 (19) | 11 (11) | 10 (11) | 5 (5)
Nasopharyngitis (Infections and infestations) | 24 (25) | 18 (18) | 22 (22) | 21 (26) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 84 (99) | 78 (88) | 72 (79) | 52 (58) | 36 (42)
Injection site tenderness (General disorders) | 58 (58) | 59 (59) | 67 (67) | 59 (59) | 18 (18)
Injection site erythema (General disorders) | 64 (64) | 63 (63) | 87 (87) | 54 (54) | 26 (26)
Injection site swelling (General disorders) | 22 (22) | 20 (20) | 21 (21) | 13 (13) | 4 (4)
Fever (General disorders) | 51 (51) | 62 (62) | 64 (64) | 48 (48) | 21 (21)
Vomiting (Gastrointestinal disorders) | 60 (60) | 57 (57) | 53 (53) | 39 (39) | 16 (16)
Crying Abnormal (Psychiatric disorders) | 58 (58) | 54 (54) | 50 (50) | 41 (41) | 21 (21)
Drowsiness (Nervous system disorders) | 58 (58) | 53 (53) | 53 (53) | 38 (38) | 20 (20)
Appetite Lost (Metabolism and nutrition disorders) | 82 (82) | 71 (71) | 74 (74) | 57 (57) | 27 (27)
Irritability (Psychiatric disorders) | 91 (91) | 79 (79) | 79 (79) | 65 (65) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.